CLINICAL TRIAL: NCT01472497
Title: Effects of Pioglitazone and Glimepiride in Hypertensive Patients - Relationship With AGE, Inflammatory Cytokines and Cardiac Markers -
Brief Title: Effects of Pioglitazone in Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tottori University Hospital (Other)
Responsible Party: Principal Investigator, Kazuhide Ogino, Associate Professor, Tottori University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PIO and HTN
Record Dates: First submitted 2011-07-21; First posted 2011-11-16 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension; Insulin Resistance
Keywords: hypertension; insulin resistance; oral glucose tolerance test; AGE; inflammatory cytokine
MeSH Terms: conditions — Hypertension; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- glymepiride (Experimental)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — pioglitazone (15mg) once a day for 24 weeks
  Other Names: actos

SUMMARY:
Insulin resistance is often complicated with hypertension. AGE and inflammation play important roles in insulin resistance. Some studies reported that pioglitazone, insulin sensitizer, is effective for patients with insulin resistance, however, the mechanisms are still unclear. The aim of this study to evaluate the effect of pioglitazone compared with glimepiride on AGE, inflammatory cytokines and cardiac markers (BNP and echo) in hypertensive patients during oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension with insulin resistance

Exclusion Criteria:

* Chronic systolic heart failure, ACS

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-04; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
advanced glycation end-product (AGE) | 24 weeks
inflammatory cytokines (TNF-alfa, IL-6 and MCP-1) | 24 weeks
cardiac function (echo and BNP) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhide Ogino, MD, Principal Investigator — Tottori University Hospital
Locations (1):
- Tottori University Hospital, Yonago, Japan